CLINICAL TRIAL: NCT02562027
Title: Objective Treatment Allocation With SBRT vs. Surgery in High Risk Patients With Early Stage Lung Cancer Within an Accountable Care Collaborative Effort Between Surgery and Radiation Oncology
Brief Title: SBRT (Stereotactic Body Radiation Therapy) vs. Surgery in High Risk Patients With Early Stage Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201509035
Record Dates: First submitted 2015-09-17; First posted 2015-09-29 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma, Non-Small-Cell-Lung; Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Aftercare; Multicenter Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-risk NSCLC participants (Experimental): * Baseline assessment of demographics and comorbidities
  * Comorbidity scoring by interview and chart review: the Adult Comorbidity Evaluation 27, Charlson Comorbidity Index, Global Initiative for Chronic Obstructive Lung Disease, Cumulative Illness Rating Scale, and COMorbidities in Chronic Obstructive Lung Disease.
  * Katz Activities of Daily Living: assessment of grip strength, walk speed, and activities of daily living
  * HRQOL questionnaires will also be administered prior to treatment and then repeated throughout follow-up: the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30, EORTC QLQ-LC13, Modified Medical Research Council, EQ-5D, CES-D, and Medical Outcomes Study Social Support Survey.
  * All questionnaire responses will be obtained with the use of a computer assisted interview system which can be used to collect data in person or through telephone interviews
  Interventions: Behavioral: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30; Behavioral: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire LC-13; Behavioral: Modified Medical Research Council; Behavioral: EQ-5D; Behavioral: Center for Epidemiological Studies Depression Scale; Behavioral: Medical Outcomes Study Social Support Survey

INTERVENTIONS:
Behavioral: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 — * 30 quality of life questions for the participant to answer
  * The first 28 questions have answers that range from 1 (Not at All) to 4 (Very Much)
  * The final 2 questions answers range from 1 (Very Poor) to 7 (Excellent)
  * Collected at baseline, 3 months post-treatment, 6 months post-treatment, 12 months post-treatment, and 24 months post-treatment
  Other Names: EORTC QLQ-C30
Behavioral: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire LC-13 — * 13 quality of life questions for the participant to answer
  * The answers range from 1 (Not at All) to 4 (Very Much)
  * Collected at baseline, 3 months post-treatment, 6 months post-treatment, 12 months post-treatment, and 24 months post-treatment
  Other Names: EORTC QLQ-LC13
Behavioral: Modified Medical Research Council — * Participants is given 5 grades to choose from ranging from 0 to 4 and participant will choose grade
  * Collected at baseline, 3 months post-treatment, 6 months post-treatment, 12 months post-treatment, and 24 months post-treatment
  Other Names: mMRC
Behavioral: EQ-5D — * 5 headings with 5 statements and the participant will check the box that best describes how he or she feels that day
  * The second part shows a scale ranging from 0 (worst health) to 100 (best health) and the participant chooses the best number on the scale
  * Collected at baseline, 3 months post-treatment, 6 months post-treatment, 12 months post-treatment, and 24 months post-treatment
  Other Names: -Collected at baseline, 3 months post-treatment, 6 months post-treatment, 12 months post-treatment, and 24 months post-treatment
Behavioral: Center for Epidemiological Studies Depression Scale — * 20 quality of life questions for the participant to answer
  * Answers range from "Rarely or none of the time" to "Most or all of the time"
  * Collected at baseline, 3 months post-treatment, 6 months post-treatment, 12 months post-treatment, and 24 months post-treatment
  Other Names: CES-D
Behavioral: Medical Outcomes Study Social Support Survey — * 19 quality of life questions for the participant to answer
  * Answers from from 1 (None of the time) to 5 (All of the time)
  * Collected at baseline, 3 months post-treatment, 6 months post-treatment, 12 months post-treatment, and 24 months post-treatment
  Other Names: MOS-SSS

SUMMARY:
A principle objective of the study is to create a validated risk model for treatment selection. This will greatly enhance the ability to counsel patients regarding their specific risks/benefit ratio for surgery or SBRT. This will improve informed decision making on the part of the patient, and remove much of the subjectivity of treatment selection.

DETAILED DESCRIPTION:
The development of SBRT for treatment of stage I NSCLC (non-small cell lung cancer) inspired the collaboration between thoracic surgery and radiation oncology and has prompted the investigators to work closely together to evaluate the relative role of SBRT and surgery. Comparative studies of these modalities have been limited in number and are often difficult to interpret due to variability in methodological issues. The productive collaboration has resulted in publication of several studies comparing SBRT and surgery utilizing propensity score based analyses to match patients from each group. However, matching on limited numbers of variables between patients ultimately selected for therapy based largely on their real or perceived comorbidity leads to significant reporting bias, and therefore methods to comprehensively assess comorbidity are necessary.

As extension of above, a very real ongoing challenge that the investigators have evaluated within clinical practice is that current guidelines defining the high risk patient are subjective and prone to physician bias. A recent secondary analysis of clinical trial inclusion criteria for SBRT underscored this bias by demonstrating that many patients that were considered inoperable were perhaps reasonable surgical candidates. Based on standard pulmonary function tests the inoperable SBRT patients had a diffusion capacity 33% higher than the high risk surgical patients in ACOSOG Z4032. Conversely, stratification of high risk surgical patients within ACOSOG Z4032 trial identified an extremely high risk subset (median DLCO% 30%, FEV1% 39%) with a 90-day 3+ adverse event rate of 48% compared to the lowest risk subset (DLCO% 69%, FEV1% 56%) with a 90-day 3+ adverse event rate of only 24%. In the absence of a clinical trial or a prospective database, there is currently no objective algorithm to guide the assignment of surgery versus SBRT.

Attempts to objectively stratify risk within the surgical population have been challenging. Risk models based on the European Thoracic Database and the Society of Thoracic Surgeons Database are not yet robust enough to guide decision-making regarding treatment assignment or classification of the very high risk surgical patient where alternative therapies may be preferable. Unfortunately, one of the current limitations to stratifying these high risk patients is that these patients are followed by physicians in independent specialties. The STS Thoracic Surgical Database does not include patients that undergo SBRT therefore it is difficult to create an inclusive algorithm for operable and inoperable patients. A principle objective of the study is to create a validated risk model for treatment selection. This will greatly enhance the ability to counsel patients regarding their specific risks/benefit ratio for surgery or SBRT. This will improve informed decision making on the part of the patient, and remove much of the subjectivity of treatment selection. Inclusion of unique metrics such as HRQOL data will further bolster the benefit to the patient by making it more patient-centric, rather than focusing on cancer outcomes alone.

As the implementation of the Affordable HealthCare Act (AHCA) continues, physicians will experience additional pressure to cut costs while maintaining or improving the quality of care provided. The current fee-for-service system is often criticized for being compartmentalized and fragmented without well-defined incentives for quality improvement.

Initiatives of the AHCA have included efforts to test care models to reduce hospital associated conditions, bundled payment plans for care improvement, and shared savings programs for accountable care organizations whereby participating providers who meet certain quality standards share in any savings achieved for the Medicare program. These are just some of the efforts designed to rein in the cost of medical care while improving the transparency and quality of care. Pilot efforts involving bundling of payments for coronary artery bypass grafting resulted in Medicare savings of $40 million with simultaneous reduced in-hospital mortality. These types of initiatives are likely to become more commonplace in the United States as efforts to create new models of care to constrain cost are introduced.

With the stimulus of these initiatives for novel systems of healthcare delivery the investigators recognized that a model of bundled payment for treatment of stage I NSCLC may not only reduce overall costs associated with treatment of stage I lung cancer but potentially improve the quality of care provided. At Washington University the investigators have taken a preemptive measure to create an accountable care organization (ACO) between the Department of Radiation Oncology and the Department of Thoracic Surgery with a focused approach on the treatment of stage I NSCLC. Important components of this collaborative effort include a bundled payment system for episodes of care involving the treatment selection, implementation, and follow up care of patients with stage I lung cancer as well as prospective assessment of quality of care measures.

The impetus for the development of this unique collaboration between radiation oncology and thoracic surgery stems from the ongoing interest in improving the quality of care for patients with early stage NSCLC. The clinical research focus has been on determining the best treatment strategies for the significant number of patients with stage I lung cancer considered medically inoperable or high risk surgical candidates. In the aging population, pulmonary insufficiency, cardiac disease, as well as other comorbidities may preclude surgery or place patients at significant risk for complications after surgery. The evolution of stereotactic body radiotherapy (SBRT) in the medically inoperable population has resulted in relatively low local recurrence rates ranging from 3-20% with favorable overall and disease-free survival in inoperable patients with Stage I NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed suspected or proven clinical stage I NSCLC (T1 or T2, N0, M0) with no prior treatment for this disease.
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Treatment selection model for high-risk early stage NSCLC patient population using comorbidity | Up to 90 days post treatment
  * Comorbidity scoring will be performed by interview and chart review including the Adult Comorbidity Evaluation 27 (ACE-27), Charlson Comorbidity Index (CCI), Global Initiative for Chronic Obstructive Lung Disease (GOLD), Cumulative Illness Rating Scale (CIRS), and COMorbidities in Chronic Obstructive Lung Disease (COMCOLD)
  * All of the comorbidity indices grade comorbidities from mild to severe. The investigators will use the data obtained from cumulative collected indices to determine the severity of patient comorbidities.
  * The data obtained from this group of patients will be compared with the previously obtained data from patients who had surgery for their stage I NSCLC.
Treatment selection model for high-risk early stage NSCLC patient population using risk indices | Up to 90 days post treatment
  * For determination of frailty, Fried's frailty criteria, a validated measurement tool which includes assessment of weight loss, exhaustion, activity level, grip strength, and walk speed. Fraility is classified using a validated score of 0-5 with patients scoring 4-5 considered frail, 2-3 considered intermediately frail, and 0-1 nonfrail.
  * Activities of daily living (Katz Activities of Daily Living) and instrumental activities of daily living (IADL) will be assessed. Both the ADL and IADL look at independence. The ADL has 6 questions/the IADL has 8 questions and the patient will receive a point for each question if he or she is considered independent. A score of 0 means the person if very dependent and very frail. A score of 6 (ADL) or 8 (IADL) means a person if very independent and not frail.
  * The data obtained from this group of patients will be compared with the previously obtained data from patients who had surgery for their stage I NSCLC.
Treatment selection model for high-risk early stage NSCLC patient population using HRQOL (health related quality of life) endpoints | Up to 24 months post treatment
  * HRQOL will be measured by the European Organization for Research and Treatment of Cancer (EORTC), Quality of Life Questionnaire (QLQ) C30, EORTC QLQ-LC13, Modified Medical Research Council (mMRC), EQ-5D, CES-D, and Medical Outcomes Study Social Support Survey (MOS-SSS).
  * Utility assessments will also be used and will serve as a quantitative measure of patient preferences and will be utilized to estimate quality adjusted life years (QALYs) to better incorporate quantity of survival, as well as quality of life consequences of stage I lung cancer interventions.

SECONDARY OUTCOMES:
Potential savings in cost using the model in this study | Up to 90 days
  Cost savings will be described with both Medicare allowable dollars and actual professional and technical costs per patient through collaboration with the Siteman Cancer Center and Barnes Jewish Hospital. Cost savings will also be reviewed with regard to pre- vs. post-ACO utilization. Cost-effectiveness analyses with regard to toxicity and quality of life will be performed using a Markov decision model and estimated with a microsimulation process
Comprehensive collaborative REDCap database to support the retrospective and prospective data collection | Up to 5 years post treatment
  * REDCap is a secure web application geared to support collection of research data
Costs of surgery | Up to 90 days
Costs of SBRT | Up to 90 days
Potential cost savings with implementation of a novel ACO for stage I NSCLC | Up to 90 days
Compare data between patients undergoing operative treatment and non-operative treatment for stage I NSCLC as measured by the combination of comorbidity, disability, and frailty indices | Up to 90 days post treatment
Quality of life indices as measured by the differences at baseline and after treatment using the implementation of the ACO | Up to 24 months post treatment
Knowledge-based treatment selection regression model for prediction of treatment-related outcomes | Up to 24 months post treatment
  This model may be used for subsequent selection of patients for operative and nonoperative therapy in patients with Stage I NSCLC based on short-term morbidity, mortality, impact on qualify of life, and cost with the potential to construct a composite outcome index based on these variables

CONTACTS AND LOCATIONS:
Overall Officials: Cliff Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu